CLINICAL TRIAL: NCT01362868
Title: Water Drinking Test (WDT) During Continuous Recording of Intraocular Pressure Fluctuation
Brief Title: Water Drinking Test During Intraocular Pressure Fluctuation (IOP) Monitoring
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too low effect on the output and low rate of responders
Sponsor: Sensimed AG (Industry)
Responsible Party: Pr. André Mermoud, Clinique de Montchoisi
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1012
Record Dates: First submitted 2011-05-27; First posted 2011-05-30 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Healthy Subjects
Keywords: Glaucoma; Triggerfish; Water drinking test
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SENSIMED Triggerfish® — Soft contact lens-based device for the continuous monitoring of IOP fluctuations

SUMMARY:
The purpose of this study is to investigate the investigational device capacity to detect an intraocular pressure increase (IOP)induced by water intake.

DETAILED DESCRIPTION:
32 subjects will be enrolled in the investigation. Eligible subjects will receive one session of 4-6-hour continuous IOP monitoring with SENSIMED Triggerfish® following water drinking test (WDT). SENSIMED Triggerfish® will be installed randomly on right or left eyes and the IOP recording will be initiated as soon as the adaptation of the device on the subject's eye is satisfying. Sensor fitting in the eye will then be evaluated every 60 minutes, until no more spontaneous Sensor movement and rotation are observed. Then IOP will be measured on the contra lateral eye using Goldmann tonometer and the subjects will be asked to drink 1 liter of water within 5 minutes.

After the water drinking, IOP will be measured on the contra lateral eye 10 minutes after the beginning of the test then every 5 minutes until returned to normal. The IOP will be measured again every 20 minutes until 2 hours after the water drinking.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer without previous ocular medical history
* 18 years or more at inclusion
* Maximal weight: 100kg
* BMI lower or equal to 30 kg/m2
* Subjects having provided informed consent

Exclusion Criteria:

* Silicone allergy
* Cardiovascular disease
* Diabetes
* Narrow or closed iridocorneal angle

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
SENSIMED Triggerfish® signal increase when Goldman IOP increase is ≥ 3 mmHg following WDT | 30-45 min after WDT

CONTACTS AND LOCATIONS:
Overall Officials: André Mermoud, MD, Principal Investigator — Clinique de Montchoisi
Locations (1):
- Unité de Glaucome, Clinique de Montchoisi, Lausanne, Switzerland